CLINICAL TRIAL: NCT06958276
Title: Changes in Shoulder Strength, Mobility, and Muscle Recruitment Following Ultrasound-Guided Percutaneous Neuromodulation in CrossFit Athletes With Nonspecific Shoulder Pain: A Randomized Controlled Trial
Brief Title: Effect of US-Guided PNM in CrossFit With Nonspecific Shoulder Pain
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Universidad de Zaragoza (Other)
Collaborators: Aragon Institute for Health Research (IIS Aragón) (Unknown)
Responsible Party: Principal Investigator, Alberto Carcasona Otal, Principal Investigator, Universidad de Zaragoza
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: NMP-e, CrossFit, dolor hombro
Record Dates: First submitted 2025-04-19; First posted 2025-05-06 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Nonspecific Shoulder Pain; Shoulder Pain Syndrome
Keywords: neuromodulation; percutaneous; ultrasound; axillary nerve; suprascapular nerve

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Masking Description: The participant will not be aware of which type of intervention they are receiving, as both interventions involve the application of a single session of US-guided PNM. The only difference between groups lies in the stimulation frequency: 10 Hz for one group and 1 Hz for the other, making it indistinguishable for the participant. Additionally, the evaluator will be different from the researcher responsible for administering the interventions and will therefore also be blinded to the type of intervention each participant has received.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- US-guided PNM 10 Hz (Experimental): One session of US-guided PNM at a frequency of 10 Hz.
  Interventions: Other: Ultrasound Guided Percutaneous Neuromodulation. Frequency of 10 Hz
- US-guided PNM 1 Hz (Experimental): One session of US-guided PNM at a frequency of 1 Hz.
  Interventions: Other: Ultrasound Guided Percutaneous Neuromodulación. Frequency of 1 Hz

INTERVENTIONS:
Other: Ultrasound Guided Percutaneous Neuromodulation. Frequency of 10 Hz — The US-guided PNM intervention will be performed with the patient in the prone position, the shoulder to be treated flexed at 90 degrees, the humerus partially supported on the table, the elbow flexed at 90 degrees, and the musculature relaxed. Needles will be inserted near the perineurium of the axillary and suprascapular nerves. Prior to needle insertion, the skin will be cleaned with isopropyl alcohol and chlorhexidine. The PNM intervention will consist of applying a compensated asymmetric biphasic current, with a rectangular positive phase and a triangular negative phase, at a frequency of 10 Hz, pulse width of 240 μs, and the maximum tolerated intensity that elicits a painless maximal muscle contraction, following this protocol: 10 stimulations of 10 seconds each, with a 10-second rest between stimulations.
  Arms: US-guided PNM 10 Hz
Other: Ultrasound Guided Percutaneous Neuromodulación. Frequency of 1 Hz — Same intervention as previously described, with the only difference being that the frequency will be 1 Hz instead of 10 Hz.
  Arms: US-guided PNM 1 Hz

SUMMARY:
CrossFit is a high-intensity physical training program that combines exercises from various disciplines, such as weightlifting, track and field, running, and gymnastics. The three main characteristics of this sport discipline are as follows: first, the execution of functional movements; second, performing them at high intensity; and lastly, constant variation. This training model has shown improvements in strength, power, balance, flexibility, and cardiorespiratory capacities.

There are various risk factors described in the literature that may lead to injuries in CrossFit athletes. It has been suggested that demanding training programs increase this risk, especially when performed incorrectly (poor technique). Additionally, excessive training load and frequency can lead to early fatigue, greater perceived effort, and risky movement execution.

On the other hand, older age, male sex, and previous injuries also appear to be relevant risk factors, as well as performing stretches prior to CrossFit practice. Several studies have shown that the shoulder is the joint with the highest prevalence of injury in this sport, surpassing other commonly affected joints such as the lumbar spine or the knee.

Among the wide variety of injuries related to the shoulder, the diagnosis of "nonspecific shoulder pain" has a high prevalence in the adult population. This term is used to describe clinical cases where it is not possible to identify the specific cause of the pain, and is justified by its multifactorial etiology, which is associated with several risk factors. These include: imbalance in the strength ratio between internal and external rotators, limitations in rotational mobility of the glenohumeral joint, deficits in motor control of the scapular musculature, shoulder muscle fatigue, and the repetitive execution of overhead exercises.

This last factor is especially relevant in the CrossFit population, as such movements are frequent in the discipline. Repeated overhead exercises have been associated with a deficit in glenohumeral internal rotation. From a biomechanical perspective, this movement is more efficient when accompanied by external rotation, so internal rotation limitation can compromise the motion. This deficit has been linked to modifiable musculoskeletal factors such as posterior capsule stiffness, shortening of the infraspinatus or teres minor muscles, and scapular mechanics alterations, as well as non-modifiable factors like bone torsion observed in young athletes. These conditions can lead to pain and/or glenoid labrum pathology.

Regarding the clinical management of nonspecific shoulder pain, conservative physiotherapy treatment is the most common approach. This is based on manual therapy and therapeutic exercise. However, in recent years, invasive physiotherapy has gained popularity in the treatment of musculoskeletal disorders through techniques such as ultrasound-guided percutaneous neuromodulation (US-guided PNM). This technique involves delivering electrical stimulation through an acupuncture needle placed near the nerve (epineurium) or the motor point of the target muscle, aiming to restore proper functionality of pathological neuromuscular structures.

US-guided PNM, applied to both the lower and upper limbs, has shown effectiveness in both healthy individuals and subjects with various musculoskeletal disorders, improving pain, strength, flexibility, and normalization of neural excitability.

Currently, there are therapeutic exercise protocols used for both evaluation and treatment of nonspecific shoulder pain in CrossFit athletes. Additionally, there are US-guided PNM protocols that have been applied to healthy CrossFit athletes and have demonstrated improvements in shoulder rotational strength. However, US-guided PNM has not yet been studied in a population of CrossFit athletes with nonspecific shoulder pain. Therefore, this randomized clinical trial aims to evaluate the effectiveness of two different US-guided PNM protocols, analyzing which methodology is most appropriate for reducing the risk factors associated with the development of nonspecific shoulder pain in CrossFit athletes.

ELIGIBILITY:
Inclusion criteria:

* Be over 18 years old.
* Have shoulder pain lasting more than 3 months.
* The pain must not have an apparent cause, meaning there is no specific diagnosis, and thus it is considered nonspecific pain.
* Train CrossFit at least 3 days per week.

Exclusion criteria:

* Have received any medical or physiotherapy treatment for nonspecific shoulder pain.
* Have had previous shoulder surgery.
* Present fear of needles (belonephobia) or fear of the US-guided PNM intervention.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2025-05-01 (Actual); Primary Completion 2025-06-01 (Actual); Study Completion 2025-07-31 (Actual)

PRIMARY OUTCOMES:
Strength ratio between ER/IR | The measurements were taken pre-intervention and immediately post-intervention.
  A hand-held dynamometer (HHD) with units in kg of force (KgF) was used. The participant was positioned according to the instructions of Hams et al., seated with the hip and knee flexed at 90 degrees, feet flat on the floor, trunk upright, shoulder at 0 degrees of abduction and neutral rotation, and elbow in contact with the trunk, flexed at 90 degrees. The dynamometer was placed on the distal third of the inner forearm to assess internal rotation (IR) and on the distal third of the outer forearm to assess external rotation (ER). Athletes were instructed to produce the maximum isometric force for 10 seconds, while the evaluator applied the same force in the opposite direction. Three tests were performed bilaterally, with a one-minute rest between each test, and the final data was the average of the three tests. The strength ratio was calculated by dividing ER/IR, with 2:3 (0.66) considered the ideal ratio.

SECONDARY OUTCOMES:
Glenohumeral rotational mobility | The measurements were taken pre-intervention and immediately post-intervention.
  A digital goniometer (HALO), which has demonstrated validity and reliability for measurements in the shoulder joint, was used. For each participant, bilateral internal rotation (IR) and external rotation (ER) were measured. Subsequently, both rotations were summed to create a third variable: the total rotational movement arc (ART). The patient was placed in the supine position, with the shoulder abducted at 90 degrees, the elbow flexed at 90 degrees, and the forearm perpendicular to the floor. An evaluator stabilized the scapula by applying pressure to the coracoid process, while another evaluator performed passive internal/external rotation and placed the goniometer on the distal third of the forearm on its dorsal side. Passive mobilization was completed when the first "end-feel" was reached or when the scapula began to move. Two measurements of each rotation were taken on each shoulder, and the final data was the average of both measurements.
Scapular motor control | The measurements were taken pre-intervention and immediately post-intervention.
  A surface electromyograph from the commercial brand Mdurance, which has been validated and used in the literature, was used. According to Kibler et al., proper scapular motor control is primarily achieved through the upper and lower trapezius muscles and the serratus anterior. Therefore, surface electrodes were placed bilaterally on the three muscles mentioned, and the athlete was asked to perform five repetitions of glenohumeral abduction in the scapular plane. The electromyograph software recorded the activation level of the three muscles, as well as the order of activation of the musculature.

CONTACTS AND LOCATIONS:
Overall Officials: Alberto Carcasona, Physiotherapist, Principal Investigator — IIS Aragón, University of Zaragoza
Locations (1):
- University of Zaragoza, Zaragoza, Zaragoza, Spain

IPD SHARING:
Plan to Share IPD: Yes
Data will be shared on a reasonable request contacting with the main author once data has been published.
  Anyway, Individual participant data (IPD) will be shared with other researchers in accordance with data sharing protocols and participant consent, ensuring confidentiality and ethical considerations are maintained.
Supporting Information: Study Protocol, SAP, ICF
Time Frame: Once research has been published
Access Criteria: Study protocol will be publish in a scientific journal